CLINICAL TRIAL: NCT02093299
Title: RIsk of Apoplexia Cerebri in CLOpidogrel Non-responders
Acronym: RISCLON
Status: Terminated | Type: Observational
Why Stopped: Lack of feasiability
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-004748-23; 2011-004748-23 (EudraCT Number)
Record Dates: First submitted 2014-03-19; First posted 2014-03-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Clopidogrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Stroke: clopidogrel 75 mg
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — a blood sample is drawn on all patients to determine responder status
  Other Names: non-responders; VeryfyNow

SUMMARY:
Stroke patients are given prophylactic treatment with clopidogrel to prevent new strokes. Some of these patients (the investigators don't know precisely how many, but previous studies indicate 4-34%) are so called non-responders, when you measure on a blood sample from the patient. These patients may have an increased risk for less effect of the treatment and therefore a higher risk for a new stroke.

The investigators want to investigate if clopidogrel non-responders have a clinically increased risk of a new stroke by following the patients for two years. With this study the investigators aim to ensure that all patients get the best prophylactic treatment and reduce the risk of early death and dependency of others.

DETAILED DESCRIPTION:
Background and purpose

Patients, who have had a stroke, have an increased risk of a new stroke. Clinical trials have proven that inhibition of blood platelets reduce the risk of a new stroke. Unfortunately there are patients not responding (non-responders) to anti-platelet treatment. Patients not responding might have a greater risk of a new stroke compared to patients responding (responders) to anti-platelet treatment.

These clinical trials does not take into account that an unknown number of the patients are unresponsive (non-responders) to inhibition of blood platelet treatment and thereby in a poorer prophylactic treatment than necessary and have a higher risk of early death, disability and depending upon others.

Trials of other anti-platelet regimes (acetylsalicylic acid) have shown that 33 % of stroke patients are non-responders and that they had an 10 times increased risk of vascular death, myocardial infarction or stroke in the first two years after the stroke and start of treatment. Therefore it is likely that it is of great clinical importance to identify non-responders to optimize therapy.

Today Clopidogrel is the drug-of-choice in prophylactic stroke treatment. To our knowledge no one has studied the non-responder problem of Clopidogrel as prophylactic treatment in stroke patients. Due to genetic differences, data from other studies can't be transferred to Danish patients.

The Clopidogrel non-responder problem has been studied in other groups of patients and they have shown that up to 34% of the patients are Clopidogrel non-responders.

This project is of great significance to the patient, their relatives and socioeconomic. The non-responder problem will be studied in a Danish population and the patients who do not respond to the drug-of-choice will receive another treatment. By this we better prevent that the patient has another stroke and thereby minimize the risk of previous death, loss of function and depending upon others.

The study is to our knowledge the first to systematically study the risk of stroke in patients in prophylactic Clopidogrel treatment who are non-responders.

The study is one of several studies with research-fellowship at Department og Neurology, Roskilde University Hospital.

Project summary Stroke patients admitted to the Stroke Unit will be included in the project. Patients who receive Clopidogrel will 2 weeks after discharge be called to the outpatient clinic and undertake a blood sample to determine whether they are Clopidogrel responders or non-responders.

The patient will be followed in the outpatient clinic every 3 months for two years by a doctor or project nurse as outpatient visits alternating phone calls to ensure that the patient follows the prescribed treatment and to determine if the patient has had a new stroke.

We estimate that 200 patients will be included in the study.

Design, recruitment, method. The study is a double blinded follow-up study of non-responders to Clopidogrel and systematic statement of healthcare data suspected of influence on the results of the study.

Patient admitted with stroke and receiving prophylactic treatment with Clopidogrel on the day of discharge will be included in the study after orally and written informed consent.

Ethics The study will follow the Helsinki Declaration of 1984, modified at the 41. World Congress in Hong Kong 1989. The study i already reported to the local Datatilsynet and approved by the local ethics committee (Region Sjællands Videnskabsetiske Komite). The study is pending approval at the Danish Medical Agency (Sundhedsstyrelsen).

Blood samples taken in the study will not delay the time to start of prophylactic treatment. Patients in the study will be treated the same as patients not included in the study.

Project benefits In Denmark 10 000 people suffer from stroke every year. Some dies almost instantly while others are disabled for life and some recover fully. These patients all have an increased risk of a new stroke.

Today the treatment of stroke is limited to a very small percentage of the patients and we know that prophylactic treatment is very important. Reducing the risk of stroke reduces the risk of early death, disability and depending upon others. The project thereby benefits the patient in the study, future stroke patients and their relatives and socio economics.

The project will be externally monitored by the Good Clinical Practice unit in Denmark and all changes to the project protocol will be reported to the local ethics committee (Region Sjællands Videnskabsetiske Komite) and the Danish Medical Agency (Sundhedsstyrelsen).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to neurological department with stroke signs om CT or MRI or history consistent with stroke and gives clopidogrel 75 mg as prophylactic treatment.

Exclusion Criteria:

* cancer diagnosis Other anti platelet treatment

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First time stroke patients
Sampling Method: Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2012-12; Primary Completion 2016-11-22 (Actual); Study Completion 2016-11-22 (Actual)

PRIMARY OUTCOMES:
Number of patient with new stroke | 2 years

SECONDARY OUTCOMES:
Number of patients with transitory ischemic attack | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Rath, MD, Principal Investigator — Dept. of Neurology Roskilde University Hospital
Locations (1):
- Neurologisk afdeling, Roskilde, Denmark